CLINICAL TRIAL: NCT05249647
Title: Effects of Instrument Based Fascial Abrasion Versus Myofascial Release Technique in Patients Having Cervicogenic Headache
Brief Title: Instrument Based Fascial Abrasion Versus Myofascial Release Technique in Cervicogenic Headache Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AH/21/0128/Warda Zafar
Record Dates: First submitted 2022-02-01; First posted 2022-02-22 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Cervicogenic Headache
Keywords: Neck and head pain
MeSH Terms: conditions — Post-Traumatic Headache; Headache | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument based fascial abrasion technique (Experimental): IASTM using tools over Myofascial trigger points of the length of targeted muscles (SCM, descending fiber of trapezius, suboccipitalis muscles) in a multidirectional stroking fashion applied to the skin at 30°- 60° for 5 minutes. Participants were in a comfortable position during treatment. Emollient (anti-allergic) was applied to prevent skin irritation prior to Fascial Abrasion application. Each session included 1 minute of sweeping (longitudinal strokes performed parallel to the muscle fibers similar to compression with oscillations) directly over the Myofascial trigger points, 2 minutes of fanning (one end of the instrument was held in place & the other end moved through a semicircular pattern similar to petrissage) and concluded with 1 min of sweeping.
  Interventions: Other: Instrument based Fascial abrasion technique
- Myofascial release technique (Active Comparator): All participants will get Conventional therapy i.e heating pad for 10 minutes. For the application of technique, the patient position will be supine lying with head fully supported on therapist hands and therapist places 3 middle fingers just inferior to the nucle line, lifts the finger tips towards the ceiling while resting the head on the table and then therapist applied a gentle upward pull. This procedure done for 2-3 minutes, 5-7 repetitions, 3 sessions per week on alternate days given for 6 weeks.
  Interventions: Other: Myofascial release technique

INTERVENTIONS:
Other: Instrument based Fascial abrasion technique — Participants were in a comfortable position during treatment. Emollient (anti-allergic) was applied to prevent skin irritation prior to Fascial Abrasion application. Each session included 1 minute of sweeping (longitudinal strokes performed parallel to the muscle fibers similar to compression with oscillations) directly over the Myofascial trigger points, 2 minutes of fanning (one end of the instrument was held in place & the other end moved through a semicircular pattern similar to petrissage) and concluded with 1 min of sweeping. Fascial Abrasion tool was washed in alcohol-based sanitizer before and after every treatment session and all norms of COVID-19 precautions were maintained. Myofascial trigger points were marked with a 1×1 cm piece of tape/under wrap to confirm consistency of subsequent treatments.
  Other Names: Instrument based soft tissue release technique
  Arms: Instrument based fascial abrasion technique
Other: Myofascial release technique — All participants will get Conventional therapy i.e heating pad for 10 minutes. For the application of technique, the patient position will be supine lying with head fully supported on therapist hands and therapist places 3 middle fingers just inferior to the nucle line, lifts the finger tips towards the ceiling while resting the head on the table and then therapist applied a gentle upward pull. This procedure done for 2-3 minutes, 5-7 repetitions, 3 sessions per week on alternate days given for 6 weeks.
  Other Names: Soft tissue release technique
  Arms: Myofascial release technique

SUMMARY:
Study will be randomized clinical trial. Data will be collected from non probability consecutive sampling technique. Total 44 participants from Rafiqa Hospital and District Headquarter (DHQ) Sargodha will be selected and randomly allocated to two different groups i.e Group A and Group B. Group A will be treated with Instrument assisted Fascial Abrasion and Conventional Therapy for 5 minutes, 6 sessions (3 sessions per week) (12) while Group B will be treated with Myofascial Release Technique and Conventional Therapy for 2 to 3 minutes, 5-7 repetitions and 3 sessions per week on alternate days were given for 6 weeks. NPRS, MOS-36, NDI will be used as outcome measuring tool before and after treatment. Data will be analyzed by using Statistical package for social sciences 25.

DETAILED DESCRIPTION:
Cervicogenic headache is a symptomatic headache characterized by chronic, hemi cranial pain syndrome in which pain sensations originates in cervical spine and soft tissues of the neck and basically referred to head. Cervicogenic headache originates in the upper cervical region, and the headache mechanism involves nociceptive structures such as the upper cervical spinal nerves, ganglia, disks, facet joints, muscles, and ligaments. Consequently, the anatomical structures innervated by cervical roots C1-C3 are potential sources of Cervicogenic headache.

Myofascial Release (MFR) is a therapeutic technique that uses gentle pressure and stretching (in both forms of direct and indirect approaches) with the intention of restoring decrease pain, optimizing length and facilitating the release of fascial restrictions caused by injury, stress, repetitive use, etc. There are some studies about MFR and its effects which include: increase extensibilities of soft tissues, increase ROM, improves joint biomechanics, increases temperature of fascia, increases blood circulation to the muscles and decreases pain and muscles tone significantly.

Although; a lot of remedies such as physiotherapy, electrotherapy, exercises therapy and spinal mobilization are used for cervicogenic headache, but sub-occipital MFR for Cervicogenic headache has not been studied specifically. Another technique used for cervicogenic headache includes Fascial Abrasion Technique tool that is a revolutionary tool that can quickly and effectively loosen muscle tissue/fascia. It improves range and quality of movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients having headaches with neck stiffness and pain.
* Headache for the past 3 months at least once per week.
* Positive flexion rotation test and restriction greater than 10°
* Patient aged 18-66 years old.

Exclusion Criteria:

* Headache not of cervical origin.
* Physiotherapy or chiropractic treatment in the past 3 months.
* Headache with autonomic involvement, dizziness and visual disturbance.
* Congenital conditions of Cervical spine

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | 6 weeks
  Scale consists of 4 questions regarding actual pain level, zero indicates no pain and 10 indicates worst pain imaginable
Neck disability index to measure functional status of neck | 6 weeks
  Scale consists of 10 sections,each section contains questions regarding head/ neck pain and some questions regarding the daily activities that we perform.
Medical outcome study( MOS-36) to measure functions of daily living | 6 weeks
  Questionnaire consists of 11 questions regarding functions of daily living

SECONDARY OUTCOMES:
Measuring tape for measuring ranges at cervical region | 6 weeks
  It is used to measure the ranges of cervical region (cervical flexion, extension, rotation and side banding)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study Principal Investigator
Locations (1):
- Warda Zafar, Sargodha, Sargodha,Punjab,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No